CLINICAL TRIAL: NCT00503906
Title: A Phase II Study of Abraxane, Avastin and Gemcitabine for First Line Metastatic Breast Cancer
Brief Title: Abraxane, Avastin, and Gemcitabine as First-Line Therapy for Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060913; SCCC-2006081 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane, Avastin and Gemcitabine (Experimental): Each treatment cycle is 28 days. Participants will be treated until disease progression:
  * Gemcitabine: 1500 mg/m2 body surface area (BSA) intravenously (IV) over 30 minutes (+/- 5 minutes) on days 1 and 15 of each cycle, followed by;
  * Abraxane: 150 mg/m2 IV over 30 minutes (+/- 5 minutes) on days 1 and 15 of each cycle, followed by;
  * Avastin: 10 mg/kg IV on days 1 and 15 of each cycle.
  Interventions: Drug: Avastin; Drug: Gemcitabine; Drug: Abraxane

INTERVENTIONS:
Drug: Avastin
  Other Names: Bevacizumab
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Abraxane
  Other Names: Albumin-Bound Paclitaxel Formulation

SUMMARY:
The investigators hypothesize that the combination of Gemzar®, Abraxane® and Avastin will increase the progression-free survival (PFS) in patients with first line metastatic breast cancer and in patients who received neoadjuvant and/or adjuvant chemotherapy present with definable metastatic disease, 6 or more months after primary treatment.

DETAILED DESCRIPTION:
This is a phase 2, single arm study. Participants will be treated with combination Gemzar, Abraxane and Avastin therapy until disease progression. Each treatment cycle is 28 days.

ELIGIBILITY:
Inclusion Criteria

1. Patients must either be:

   * treatment-naïve with newly diagnosed her2neu non-overexpressing (non amplified) metastatic (Stage IV) breast cancer, or
   * HER2/neu-negative patients with metastasis diagnosed 6 or more months after completing primary systemic treatment (neoadjuvant, adjuvant chemotherapy).
2. No previous chemotherapy regimen for metastatic breast cancer.
3. 18 years of age or older.
4. Measurable disease as defined by RECIST criteria or evaluable disease.
5. Eastern Cooperative Oncology Group (ECOG) 0-1.
6. Life expectancy greater than 3 months.
7. For female (or male) patients, either pre- or post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control for the duration of the study
8. Provide written informed consent before any study-related procedure not part of normal medical care is conducted
9. Willing and able to comply with the protocol requirement
10. Laboratory parameters as follows:

    * Neutrophils: 1.5 x109/L or greater
    * Platelets: 100 x109/L or greater
    * Hemoglobin: ≥ 9.0 g/dL
    * Serum Creatinine: ≤ 1.5mg/dL
    * Bilirubin: ≤ ULN, except when caused by metastatic disease
    * Alanine transaminase (ALT)/Aspartate transaminase (AST): ≤ 2.5 times the upper limit of the normal range (ULN) except when caused by metastatic disease
    * Urine protein creatinine (UPC) ratio < 1.0 at screening.

Exclusion Criteria

1. Previous treatment with gemcitabine.
2. History of Gastrointestinal Bleeding in the previous 3 months.
3. Chemotherapy within 4 weeks prior to enrollment.
4. Radiation therapy or evidence of acute effects of radiation therapy within 2 weeks prior to enrollment.
5. Any major surgery within 4 weeks prior to enrollment.
6. Presence of central nervous system or brain metastases.
7. Urine protein: creatinine ratio ≥ 1.0 at screening.
8. Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
9. A prior history of hypertensive crisis or hypertensive encephalopathy.
10. Peripheral neuropathy > grade I.
11. Clinical AIDS or known positive HIV serology
12. No concurrent clinically evident malignancy is allowed except inactive non-melanoma skin cancer and inactive cervical cancer diagnosed or other cancer for which the patient has been disease-free for five years.
13. Unstable angina.
14. New York Heart Association (NYHA) Grade II or greater congestive heart failure
15. History of myocardial infarction within 6 months.
16. History of stroke within 6 months.
17. Clinically significant peripheral vascular disease.
18. Evidence of bleeding diathesis or coagulopathy
19. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, anticipation of need for major surgical procedure during the course of the study.
20. Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to enrollment.
21. Pregnant (positive pregnancy test) or lactating.
22. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to enrollment
23. Serious, non-healing wound, ulcer, or bone fracture
24. Inability to comply with study and/or follow-up procedures
25. Participants with serious medical or psychiatric illness that would render chemotherapy unsafe are ineligible.
26. Participants cannot have been in another experimental drug study other than a Bevacizumab cancer study within 4 weeks of the first infusion of these study medications.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Glück, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Result] Lobo C, Lopes G, Baez O, Castrellon A, Ferrell A, Higgins C, Hurley E, Hurley J, Reis I, Richman S, Seo P, Silva O, Slingerland J, Tukia K, Welsh C, Gluck S. Final results of a phase II study of nab-paclitaxel, bevacizumab, and gemcitabine as first-line therapy for patients with HER2-negative metastatic breast cancer. Breast Cancer Res Treat. 2010 Sep;123(2):427-35. doi: 10.1007/s10549-010-1002-0. Epub 2010 Jun 29. PMID 20585851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abraxane, Avastin and Gemcitabine
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.2)
Age, Continuous [Median (Full Range); unit: years] | 53.8 [34 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival
Description: Progression-free survival will be measured from the first dose date to the earliest date of documented evidence of progressive disease or the date of death due to any causes, whichever occurs first.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 29
months | 10.4 [5.6 to 15.2]

2. Secondary Outcome: Rates of Partial Response (PR), Complete Response (CR) and Overall Response (ORR) in Study Participants
Description: Rates of partial response (PR), complete response (CR) and overall response (PR+CR = ORR) in study participants according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0.
Time Frame: After two cycles, about 60 days
Population: Evaluable patients are study-eligible patients who receive an initial infusion of combination chemotherapy consisting of Gemcitabine, NAB paclitaxel and Bevacizumab and have had at least one CT scan for evaluation of disease status.
Measure: Number; unit: percentage of participants
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 29
percentage of participants
  Overall Response Rate (ORR) | 75.6
  Complete Response (CR) | 27.6
  Partial Response (PR) | 48.3

3. Secondary Outcome: Rate of Toxicity in Study Participants
Description: Determination of safety and side effect profile of the protocol therapy including the rate of toxicity in study participants. The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for adverse event reporting.
Time Frame: Over the course of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 29
percentage of participants
  Alopecia, Grade 1/2 | 65.5
  Fatigue, Grade 1/2 | 37.9
  Bone Pain, Grade 1/2 | 31
  Nausea, Grade 1/2 | 31
  Skin rash/lesions, Grade 1/2 | 27.6
  Neutropenia, Grade 1/2 | 10.3
  Grade 3/4 Toxicities | 27.6

4. Secondary Outcome: Relationship Between Circulating Tumor Cells (CTC) and Disease Progression as Measured by Presence of CTC at Baseline and Over the Course of Study Treatment
Description: Exploration of the relationship between circulating tumor cells (CTC) and disease progression, by measuring CTC at baseline and over the course of treatment.
Time Frame: Baseline, over the course of Treatment, about 1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Relationship Between SPARC Expression and Response to Protocol Therapy.
Description: Relationship between SPARC expression and response to this chemotherapy combination and relation to progression free survival.
Time Frame: Baseline, over the course of treatment, about 1 year
Population: Data were not collected for this outcome measure.
Groups:
- Abraxane, Avastin and Gemcitabine: Each treatment cycle is 28 days. Participants will be treated until disease progression:
  * Gemcitabine: 1500 mg/m2 body surface area (BSA) intravenously (IV) over 30 minutes (+/- 5 minutes) on days 1 and 15 of each cycle, followed by;
  * Abraxane: 150 mg/m2 IV over 30 minutes (+/- 5 minutes) on days 1 and 15 of each cycle, followed by;
  * Avastin: 10 mg/kg IV on days 1 and 15 of each cycle.
  Avastin
  Gemcitabine
  Abraxane
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 0

6. Post Hoc Outcome: Rate of Overall Survival in Study Participants
Description: Rate of overall survival in study participants. Overall survival will be measured from the date of enrollment to the date of death from any cause, or the date of last contact (censored observations.)
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abraxane, Avastin and Gemcitabine
Number analyzed (Participants) | 29
percentage of participants | 77.2 [51.1 to 90.5]

ADVERSE EVENTS:
Arm/Group | Abraxane, Avastin and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Avastin and Gemcitabine (N=29)
Leukopenia (Blood and lymphatic system disorders) | 1 — Grade 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 — Grade 3
Peripheral Neuropathy (Nervous system disorders) | 1 — Grade 3
PortAcath infection (Skin and subcutaneous tissue disorders) | 2 — Grade 3
Abscess (Infections and infestations) | 1 — Grade 3
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
Breast Abscess (Infections and infestations) | 1
Fever/Sepsis (Infections and infestations) | 1 — Grade 3
Hematuria (Renal and urinary disorders) | 1 — Grade 3
Neutropenic Fever (Infections and infestations) | 1 — Grade 4
Seizure/Syncope (Nervous system disorders) | 1 — Grade 3
Tamponade (Surgical and medical procedures) | 1
UTI (Renal and urinary disorders) | 1 — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Avastin and Gemcitabine (N=29)
Neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 19
Fatigue (General disorders) | 11
Bone Pain (Musculoskeletal and connective tissue disorders) | 9
Nausea (Gastrointestinal disorders) | 8
Skin rash/lesion (Skin and subcutaneous tissue disorders) | 8
Hand/Foot syndrome (Musculoskeletal and connective tissue disorders) | 7
Headache (General disorders) | 7
Epistaxis (Vascular disorders) | 6
Peripheral Neuropathy (Nervous system disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Insomnia (General disorders) | 4
Anxiety (Psychiatric disorders) | 3
Hypertension (Vascular disorders) | 3
PortAcath Disorder (Skin and subcutaneous tissue disorders) | 1
Abscess (Infections and infestations) | 1
Amenorrhea (Reproductive system and breast disorders) | 2
Blurred Vision (Eye disorders) | 2
Cough (General disorders) | 2
Depression (Psychiatric disorders) | 2
Dysgeusia (Metabolism and nutrition disorders) | 2
Flu-like symptoms (Infections and infestations) | 2
Loss of appetite (Metabolism and nutrition disorders) | 2
Lymphedema (Blood and lymphatic system disorders) | 2
Oral infection (Infections and infestations) | 2
Rhinorrhea (Infections and infestations) | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 2
Weight Loss (General disorders) | 2
Acute renal insufficiency (Renal and urinary disorders) | 1
Chest Pain (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Heat intolerance (Endocrine disorders) | 1
Hot flashes (Endocrine disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Mucositis (Infections and infestations) | 1
Painful edema (Infections and infestations) | 1
Pedal edema (Infections and infestations) | 1
Pelvic pain (General disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Reflux (Gastrointestinal disorders) | 1
Regurgitation (valve) (Gastrointestinal disorders) | 1
Scotoma (Eye disorders) | 1
Tachycardia (Cardiac disorders) | 1
Thrombus (Vascular disorders) | 1
Tricuspid Regurg (Cardiac disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes